CLINICAL TRIAL: NCT01375959
Title: The Effect of Resveratrol in Older Adults With Impaired Glucose Tolerance: a Double-Blind Crossover Study
Brief Title: Pilot Study of Resveratrol in Older Adults With Impaired Glucose Tolerance
Acronym: RSV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Jill Crandall, Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-398
Record Dates: First submitted 2011-05-12; First posted 2011-06-20 (Estimated); Results first posted 2020-08-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-09

CONDITIONS: Impaired Glucose Tolerance
Keywords: resveratrol; glucose intolerance; insulin resistance; endothelial function
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resveratrol (Experimental): resveratrol 500 mg capsules, 3 each day for 6 weeks
  Interventions: Dietary Supplement: resveratrol
- Placebo (Placebo Comparator): matching placebo capsule containing lactose, 3 each day for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: resveratrol — resveratrol 500 mg capsules, 3 capsules (1500 mg) orally twice a day for 6 weeks
  Other Names: RevGenetics; X500 Resveratrol
  Arms: Resveratrol
Drug: Placebo — 3 placebo capsules orally twice a day for 6 weeks
  Arms: Placebo

SUMMARY:
Resveratrol is a substance found in many plants, including grapes and red wine, which is widely used as a nutritional supplement. Studies in cells and lower animals show that resveratrol has many potential benefits, including prolonging lifespan, preventing cancer and heart disease and normalization of glucose metabolism. Although use of this agent shows great promise in the treatment and/or prevention of diabetes, there have been no studies reported to date in humans. As an initial step, this proposal is for a 6 week pilot study of resveratrol treatment in older adults with impaired glucose tolerance (IGT) in order to explore its effects on post-meal blood glucose metabolism. Preliminary studies will also be conducted to explore how resveratrol works by studying cellular function (in muscle samples obtained from study participants) and by testing resveratrol's effect on blood vessel function.

DETAILED DESCRIPTION:
A. Introduction and Specific Aims Resveratrol (RSV), a plant-derived polyphenol and potential activator of the mammalian sirtuin, Sirt1, has demonstrated promising effects on insulin secretion, insulin sensitivity and glucose tolerance and has extended the lifespan of obese mice. RSV is in common use as a nutritional supplement, but formal studies in humans are limited and-in particular-the metabolic effects of RSV in humans have yet to be carefully tested. The convergence of a worldwide epidemic of diabetes combined with a marked increase in the proportion of the elderly underscore the need to develop new approaches to improve glucose intolerance. We therefore propose a study of RSV treatment in older subjects with impaired glucose tolerance (IGT) to determine if there is improvement in glucose tolerance and markers of insulin resistance, mitochondrial biogenesis and vascular function. This proposal builds on our findings in a recently-completed NIH P01 on cardiovascular disease markers in older adults with IGT. It is our hypothesis that RSV has the potential to exert important metabolic effects that can be directly and safely tested in human subjects. The growing body of pre-clinical evidence, as well as our own preliminary data, provide strong support for formal tests of RSV effects on several important metabolic parameters. These proposed studies constitute a critical step in investigating the therapeutic potential of RSV, as well as providing insight into relevant mechanisms.

Specific Aims: We propose a 6-week randomized, double-blind, placebo controlled cross-over study of RSV in older adults (age 50-80 years, n=38) with IGT, with the following aims:

Specific Aim 1: To assess the effects of RSV (2g/day) on mixed meal tolerance in subjects with age-related glucose intolerance. In our previous studies, we developed a standard mixed meal protocol to evaluate postprandial changes in glucose, insulin and lipids. We will apply this protocol to study a cohort of older adults with impaired glucose tolerance in a double-blind, placebo controlled cross-over study of RSV treatment. Metabolic outcomes will include post-meal glucose area under the curve (AUC), calculated estimates of insulin sensitivity and insulin secretion and circulating levels of free fatty acids and triglycerides. This study will be the first to document RSV effects on glucose intolerance in humans and will provide critical information needed to inform future clinical and mechanistic investigations. We hypothesize that treatment with RSV will result in improvement in mixed meal tolerance, via effects on insulin secretion, insulin action or both, in subjects with age-related glucose intolerance.

Specific Aim 2: To assess the effects of RSV on age-related decline in mitochondrial biogenesis. In animal models, RSV has been shown to enhance mitochondrial biogenesis, which may occur through activation of Sirt1, which is an important regulator of cellular energy metabolism via PGC-1α (peroxisome-proliferator-activated receptor-γ coactivator-1 alpha). We will assess this directly by measuring mitochondrial mRNA expression and DNA copy number in muscle obtained from participants after treatment with RSV compared with placebo. Studies of mitochondrial morphology and enzyme activity will be performed in collaboration with Dr. Sreekumaran Nair (Mayo Clinic), who is an expert in mitochondrial physiology. We hypothesize that treatment with RSV will result in improvement in mitochondrial number and function, which is a potential mechanism for improvement in insulin sensitivity that may occur with RSV treatment.

Specific Aim 3: To assess the effects of RSV on fasting and post-meal endothelial function. Since treatment with RSV has also been reported to have beneficial cardiovascular effects, including improved vascular reactivity, we will study in vivo endothelial function. We will use reactive hyperemia peripheral arterial tonometry to assess endothelial dependent vasodilation in study subjects before and after treatment with RSV, in both the fasting and postprandial state. Augmentation index, a measure of arterial stiffness will also be assessed. We hypothesize that chronic treatment with RSV will result in improvement in endothelial function through direct vascular effects, which may be mediated via enhanced nitric oxide availability, reduced oxidative stress and/or as a consequence of improvement in glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* impaired glucose tolerance

Exclusion Criteria:

* history of estrogen-dependent neoplasm
* use of certain drugs: high dose statins, warfarin, antiepileptics
* current treatment with anti-diabetes medications
* impaired liver or kidney function

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Crandall, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine of Yeshiva University, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Resveratrol First, Then Placebo: resveratrol 500 mg capsules, 3 capsules (1500 mg) orally twice a day for 6 weeks
  wash-out period for 2 weeks
  matching placebo capsule containing lactose, 3 orally twice a day for 6 weeks
- Placebo First, Then Resveratrol: matching placebo capsule containing lactose, 3 orally twice a day for 6 weeks
  wash-out period for 2 weeks
  resveratrol 500 mg capsules, 3 capsules (1500 mg) orally twice a day for 6 weeks
Period: First Intervention (6 Weeks)
Arm/Group | Resveratrol First, Then Placebo | Placebo First, Then Resveratrol
Started | 17 | 21
Received Invertention | 17 | 21
Completed | 15 (Two participants were withdrawn due to adverse events.) | 18 (Three participants were withdrawn due to adverse events.)
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 3
Period: Wash-Out (3 Weeks)
Arm/Group | Resveratrol First, Then Placebo | Placebo First, Then Resveratrol
Started | 15 | 18
Completed | 15 | 18
Not Completed | 0 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Resveratrol First, Then Placebo | Placebo First, Then Resveratrol
Started | 15 | 18
Completed | 15 | 15
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Resveratrol First: resveratrol 500 mg capsules, 3 each day for 6 weeks
  resveratrol: resveratrol 500 mg capsules, 3 capsules (1500 mg) orally twice a day for 6 weeks
- Placebo First: matching placebo capsule containing lactose, 3 each day for 6 weeks
  Placebo: 3 placebo capsules orally twice a day for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Resveratrol First | Placebo First | Total
Number analyzed (Participants) | 17 | 21 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (8) | 67 (6) | 67 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 11 | 14 | 25
Region of Enrollment [Number; unit: participants]
  United States | 17 | 21 | 38

OUTCOME MEASURES:

1. Primary Outcome: Post Meal Glucose Area Under the Curve
Description: Glucose AUC following a standard mixed meal challenge AUC, Area Under a Curve. There are no "normal ranges" but a higher value is worse than a lower value.
Time Frame: end of each of two 6 week treatment periods
Population: Out of 38 total randomized, 35 actually received resveratrol and 36 actually received placebo.
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Groups:
- Resveratrol: Participants received resveratrol 500 mg capsules, 3 capsules (1500 mg) orally twice a day for 6 weeks.
- Placebo: Participants received placebo, 3 capsules (matching placebo capsule containing lactose), orally twice a day for 6 weeks.
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 35 | 36
mg*hr/dL | 508 (88) | 513 (80)

2. Secondary Outcome: Insulin Sensitivity Using a Modification of the Matsuda Index
Description: Insulin sensitivity was measured from insulin and glucose levels obtained following standard meal challenge using a modification of the Matsuda index. This was calculated based on data obtained from a 75 g oral glucose tolerance test, as follows: 10,000 divided by the square root of {(fasting plasma glucose X fasting plasma insulin) (mean plasma glucose X mean plasma insulin)}. This is a unitless measure.
  The Matsuda index is considered an early biomarker for metabolic dysregulation and is an effective clinical tool to define insulin sensitivity (i.e., the ability of tissues to respond to the signal of insulin) and secretory defects in individuals with impaired glucose homeostasis. The Matsuda index correlates strongly with the euglycemic insulin clamp which is a direct measure of insulin sensitivity. In the United States, it is recognized that participants who do not have insulin resistance have Matsuda Index values of >=2.5.
Time Frame: end of each of two 6 week treatment periods
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 2.3 (1.7) | 2.0 (1.0)

3. Other Pre Specified Outcome: Insulin Secretion
Description: c-peptide deconvolution; HOMA-B
Time Frame: end of each of two 6 week treatment periods
Measure: Mean (Standard Deviation); unit: pmol/kg/min
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 30 | 30
pmol/kg/min | 8.9 (3.0) | 8.1 (2.5)

4. Other Pre Specified Outcome: Peripheral Microvascular Endothelial Function Via Reactive Hyperemia-Peripheral Arterial Tonometry (RH-PAT) Index
Description: Reactive Hyperemia-Peripheral Arterial Tonometry (RH-PAT) index is the ratio of the average pulse amplitude in the posthyperemic phase divided by the average baseline amplitude, with normalization to the signal in the control arm to compensate for any systemic changes. RH-PAT is a non-invasive and user-independent technique used to assess peripheral microvascular endothelial function by measuring changes in digital pulse volume during reactive hyperemia. Lower RH-PAT scores are associated with flow mediated dilatation (FMD) and may predict mortality in subjects with cardiovascular (CV) risk factors including obesity, total/HDL cholesterol ratio, diabetes, smoking and dyslipidemia.
Time Frame: end of each of two 6 week treatment periods
Measure: Mean (Standard Deviation); unit: RH-PAT Index
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 30 | 30
RH-PAT Index | 2.02 (0.2) | 1.76 (0.02)

5. Other Pre Specified Outcome: Number of Differentially Expressed Transcripts
Description: Gene expression in skeletal muscle using RNASeq
Time Frame: end of each of two 6 week treatment periods
Measure: Number; unit: differentially expressed transcripts
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 30 | 30
differentially expressed transcripts | 140 | 0

ADVERSE EVENTS:
Time Frame: During full 16 week study period
Groups:
- Placebo: matching placebo capsule containing lactose, 3 orally twice a day for 6 weeks
Arm/Group | Resveratrol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/38
Other Adverse Events (participants affected / at risk) | 8/38 | 8/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resveratrol (N=38) | Placebo (N=38)
pneumonia (Infections and infestations) | 0 (0) | 1 (1) — hospitalized for bronchitis and pneumonia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resveratrol (N=38) | Placebo (N=38)
rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
abnormal liver function (Hepatobiliary disorders) | 0 (0) | 1 (1)
abnormal electrocardiogram (Cardiac disorders) | 0 (0) | 2 (2)
elevated PSA (Renal and urinary disorders) | 1 (1) | 0 (0)
gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
weight loss (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No